CLINICAL TRIAL: NCT06210828
Title: Effectiveness of Telerehabilitation in Balance Training Program Among Elderly at Risk of Falling, a Randomized Controlled Trial
Brief Title: Effectiveness of Telerehabilitation in Balance Training Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Intouch Amphaiphan, Intouch Amphaiphan, MD, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 339/2566(IRB3)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Postural Balance; Fall
Keywords: Physical Performance; Falling; Elderly; Telerehabilitation; Telerehab; Telemedicine; Exercise; Telehealth
MeSH Terms: conditions — Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): A telerehabilitation group participates in two weekly exercise sessions over a 12-week period at home. These sessions, led by a physical therapist through two-way communication, focus on lower extremity strengthening and balance exercises. In addition to the guided sessions, participants are encouraged to perform self-directed exercises one day per week.
  Interventions: Behavioral: Telerehabilitation
- Control Group (Active Comparator): * Receive fall prevention exercise brochure that includes instructions on how to perform the exercises, the recommended repetition and number of sets.
  * Participants are suggested to perform self-directed exercises three day per week.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Telerehabilitation — Two weekly exercise sessions over a 12-week period at home via LINE Video call with physical therapist. Focusing on lower extremity strengthening and balance exercises. In addition to the guided sessions, participants are encouraged to perform self-directed exercises one day per week.
  Arms: Telerehabilitation Group
Behavioral: Control — Receive fall prevention exercise brochure
  Arms: Control Group

SUMMARY:
* The purpose of this study is to assess the effectiveness of telerehabilitation for fall prevention.
* Participants are randomly assigned to telerehabilitation group or control group.
* Both the telerehabilitation and control groups will receive fall prevention education.
* In addition, both groups will receive a fall prevention exercise brochure that includes instructions on how to perform the exercises, the recommended repetition and number of sets.
* The telerehabilitation group engages in two exercise sessions per week for a duration of 12 weeks at home. The session will be led by a physical therapist via telerehabilitation (LINE video call).
* All participants are advised to perform exercise for a total 3 days/week and record in the log book.
* Participants are evaluated for balancing abilities using tests including: Timed Up and Go test, Five times chair stand, Single leg stance, Gait speed, Number of fall at 3 month, 6 month, 1 year.

DETAILED DESCRIPTION:
* The investigators distribute invitation flyers for enrollment throughout Siriraj Hospital. Participants who comply with the eligibility criteria, can contact the researcher or outpatient clinic rehabilitation nurse to schedule an appointment.
* When a patient is willing to participate in the research, the researcher will provide the consent form for the participant to sign.
* After participants sign the informed consent, demographic data including age, sex, body weight, height, BMI, living status, educational status, functional status, gait aid use, underlying diseases, fall history, drug use, cognitive function and home environment. Baseline physical performance including Timed Up and Go test, five times chair stand, Single leg stance and gait speed are also recorded in case record form at outpatient clinic rehabilitation by an assessor who are blinded to group allocation.
* Participants are randomly assigned to telerehabilitation groups or control group with a simple randomization with a ratio of 1:1. Generate random sequence lists by an investigator who is not involved in data collection or administering interventions. The sequence generation lists are then concealed by using opaque-sealed envelopes.

Both the telerehabilitation and control groups will receive fall prevention education from a doctor after participation and checking during visiting at the outpatient clinic (the first visit, and then at 3 months, 6 months, and 1 year).

* In addition, both groups will receive a fall prevention exercise brochure that includes instructions on how to perform the exercises, the recommended repetition and number of sets.
* The telerehabilitation group engages in two exercise sessions per week for a duration of 12 weeks at home. The session will be led by a physical therapist via two way communication telerehabilitation (LINE video call). The physical therapist will record each session participated.
* Each session starts with a 10 minute warm-up, followed by 40 minutes of strengthening and balance training and ending with 10 minutes cool-down. The exercise program consists of two levels. After completing the first level for a month, participants will progress to the second level.
* Level 1 involved various exercises included: strengthening exercise emphasizing standing hip abductors; standing hip extensors; standing knee extensor; heel rise and balance exercise including sit to stand; marching, triangle step, side way walks.
* Level 2 increase in intensity of training by use an elastic band on the lower extremities during strengthening exercises. Additionally, to enhance the difficulty of balance training, reducing hand support are perform during balance exercise. The investigators will be recruiting 1-3 participants for a group of telerehabilitation.
* All participants are advised to perform exercise for a total 3 days/week and record in the log book
* Participants are evaluated for balancing abilities using tests including: Timed Up and Go test, Five times chair stand, Single leg stance, Gait speed, Number of fall at 3 month, 6 month, 1 year.
* All of the tests are conducted sequentially at baseline, after 3 months, 6 months, 1 years by an assessor who are blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly aged ≥ 60 years walking independently with or without gait aid use
2. Had a history of falling at least 1 time within the past year.
3. Participants or their caregivers have an ability to use telemedicine (LINE video call), read and understand a brochure.

Exclusion Criteria:

Those who have unstable medical conditions influenced their gait and mobility such unstable cardiopulmonary problem, non-heal fracture and severe arthritis and a cognitive impairment limited learning ability to exercise will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go test | 1 year
  time taken to rise from a chair, walk a 3-meter distance, turn around, walk back and sit down

SECONDARY OUTCOMES:
Five times chair stand | 1 year
  subjects will be asked to rise from a standard height chair five times, as fast as possible and time-spent will be recorded, as the time from the initial seated position to the final seated position after completing five stands
Single leg stance | 1 year
  subjects will be asked to stand on one leg as long as possible. The time obtained will be recorded
Gait speed | 1 year
  time taken to walk at comfortable speed over a distance of 10 meters

CONTACTS AND LOCATIONS:
Overall Officials: INTOUCH AMPHAIPHAN, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of medicine, Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark RD, Lord SR, Webster IW. Clinical parameters associated with falls in an elderly population. Gerontology. 1993;39(2):117-23. doi: 10.1159/000213521. PMID 8514201
- [Background] Sherrington C, Michaleff ZA, Fairhall N, Paul SS, Tiedemann A, Whitney J, Cumming RG, Herbert RD, Close JCT, Lord SR. Exercise to prevent falls in older adults: an updated systematic review and meta-analysis. Br J Sports Med. 2017 Dec;51(24):1750-1758. doi: 10.1136/bjsports-2016-096547. Epub 2016 Oct 4. PMID 27707740
- [Background] Gardner MM, Buchner DM, Robertson MC, Campbell AJ. Practical implementation of an exercise-based falls prevention programme. Age Ageing. 2001 Jan;30(1):77-83. doi: 10.1093/ageing/30.1.77. PMID 11322678
- [Background] Kwak CJ, Kim YL, Lee SM. Effects of elastic-band resistance exercise on balance, mobility and gait function, flexibility and fall efficacy in elderly people. J Phys Ther Sci. 2016 Nov;28(11):3189-3196. doi: 10.1589/jpts.28.3189. Epub 2016 Nov 29. PMID 27942147
- [Background] Kuptniratsaikul V, Praditsuwan R, Assantachai P, Ploypetch T, Udompunturak S, Pooliam J. Effectiveness of simple balancing training program in elderly patients with history of frequent falls. Clin Interv Aging. 2011;6:111-7. doi: 10.2147/CIA.S17851. Epub 2011 May 6. PMID 21594001
- [Background] Zhuang J, Huang L, Wu Y, Zhang Y. The effectiveness of a combined exercise intervention on physical fitness factors related to falls in community-dwelling older adults. Clin Interv Aging. 2014;9:131-40. doi: 10.2147/CIA.S56682. Epub 2014 Jan 10. PMID 24453483
- [Background] Leslie S, Tan J, McRae PJ, O'leary SP, Adsett JA. The Effectiveness of Exercise Interventions Supported by Telerehabilitation For Recently Hospitalized Adult Medical Patients: A Systematic Review. Int J Telerehabil. 2021 Dec 16;13(2):e6356. doi: 10.5195/ijt.2021.6356. eCollection 2021. PMID 35646230
- [Background] Chen JJ, Cooper DM, Haddad F, Sladkey A, Nussbaum E, Radom-Aizik S. Tele-Exercise as a Promising Tool to Promote Exercise in Children With Cystic Fibrosis. Front Public Health. 2018 Sep 28;6:269. doi: 10.3389/fpubh.2018.00269. eCollection 2018. PMID 30324099
- [Background] Peretti A, Amenta F, Tayebati SK, Nittari G, Mahdi SS. Telerehabilitation: Review of the State-of-the-Art and Areas of Application. JMIR Rehabil Assist Technol. 2017 Jul 21;4(2):e7. doi: 10.2196/rehab.7511. PMID 28733271
- [Background] Bernocchi P, Giordano A, Pintavalle G, Galli T, Ballini Spoglia E, Baratti D, Scalvini S. Feasibility and Clinical Efficacy of a Multidisciplinary Home-Telehealth Program to Prevent Falls in Older Adults: A Randomized Controlled Trial. J Am Med Dir Assoc. 2019 Mar;20(3):340-346. doi: 10.1016/j.jamda.2018.09.003. Epub 2018 Oct 23. PMID 30366759
- [Background] Ranaweera AD, Fonseka P, PattiyaArachchi A, Siribaddana SH. Incidence and risk factors of falls among the elderly in the District of Colombo. Ceylon Med J. 2013 Sep;58(3):100-6. doi: 10.4038/cmj.v58i3.5080. PMID 24081169
- [Background] Barry E, Galvin R, Keogh C, Horgan F, Fahey T. Is the Timed Up and Go test a useful predictor of risk of falls in community dwelling older adults: a systematic review and meta-analysis. BMC Geriatr. 2014 Feb 1;14:14. doi: 10.1186/1471-2318-14-14. PMID 24484314
- [Background] Tiedemann A, Shimada H, Sherrington C, Murray S, Lord S. The comparative ability of eight functional mobility tests for predicting falls in community-dwelling older people. Age Ageing. 2008 Jul;37(4):430-5. doi: 10.1093/ageing/afn100. Epub 2008 May 16. PMID 18487264
- [Background] Chang CJ, Chang YS, Yang SW. Using single leg standing time to predict the fall risk in elderly. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:7456-8. doi: 10.1109/EMBC.2013.6611282. PMID 24111469
- [Background] Hong C. Gait Speed Cut-Off Point as a Predictor of Fall in Community-Dwelling Older Adults: Three-Year Prospective Finding from Living Profiles of Elderly People Surveys in Korea. KJFP 2016;6:105-110.
- [Background] Kis O, Buch A, Stern N, Moran DS. Minimally supervised home-based resistance training and muscle function in older adults: A meta-analysis. Arch Gerontol Geriatr. 2019 Sep-Oct;84:103909. doi: 10.1016/j.archger.2019.103909. Epub 2019 Jul 8. PMID 31301519
- [Background] Ninlerd C, Dungkong S, Phuangphay G, Amornsupak C, Narkbunnam R. Effect of home-based rehabilitation exercise program for elderly patients with femoral neck fracture after bipolar hemiarthroplasty. Siriraj Med J. 2020; 72(4): 307-14
- See also: SITUATION OF 2020 THE THAI OLDER PERSONS — https://www.dop.go.th/download/knowledge/th1635826412-975_0.pdf
- See also: Falls — http://www.who.int/news-room/fact-sheets/detail/falls
- See also: Telehealth Guidelines — https://australian.physio/sites/default/files/APATelehealthGuidelinesCOVID190420FA.pdf